CLINICAL TRIAL: NCT02288403
Title: Effects of a High-intensity Interval Training Program Compared to a Moderate Intensity Program in Adults 18-44 Years
Brief Title: Interval Versus Continuous Training in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Victor Hugo Arboleda Serna, Associate Professor, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIIT-1-UdeA
Record Dates: First submitted 2014-11-04; First posted 2014-11-11 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Volunteers
Keywords: Aerobic Exercise; Oxygen Consumption; Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic interval training (Experimental): Interval exercise at an intensity between 90-95% of maximum heart rate (15x30 s), with recoveries at an equivalent speed to 50-55 % of maximal oxygen consumption at baseline (14x60 s).
  24 training sessions, 3x weekly (on alternate days).
  Interventions: Behavioral: Aerobic interval training
- Continuous training (Active Comparator): 40 minutes of continuous exercise at an intensity between 65-75% of maximum heart rate.
  24 training sessions, 3x weekly (on alternate days).
  Interventions: Behavioral: Continuous training

INTERVENTIONS:
Behavioral: Aerobic interval training
  Arms: Aerobic interval training
Behavioral: Continuous training
  Arms: Continuous training

SUMMARY:
Aerobic exercise produces increases in cardiorespiratory fitness (CF), which constitute a protective factor for cardiovascular disease and all-cause mortality. Therefore, aerobic exercise is a key strategy to promoting cardiovascular. There is some evidence that aerobic high intensity interval training may lead to greater increases in CF compared with continuous moderate-intensity training.

The main objective of this study is to examine the effects of an aerobic high intensity training program versus a continuous moderate intensity training program on CF in men 18 to 44 years.

DETAILED DESCRIPTION:
Forty-four individuals will be randomly assigned to one of two aerobic training programs on a treadmill. Both groups will performed three times a week for eight-weeks (on alternate days). Half will run 40 minutes of continuous exercise at an intensity between 65-75% of maximum heart rate, and the remaining 22 will complete 21.5 minutes of interval exercise at an intensity between 90-95% of maximum heart rate, with recoveries between 50-55 % of maximum heart rate. After each session both groups will complete eight strength exercises mainly including large muscle groups for two sets and 8-12 repetitions at an intensity equivalent to 60-70% of one repetition maximum (controlled by perceived effort). Rest between sets will be kept between 60 and 90 seconds.

All participants will be evaluated at the start and completion of the intervention for their maximal oxygen consumption, blood pressure, waist circumference, BMI, body composition, and steps per week.

ELIGIBILITY:
Inclusion Criteria:

* Perform aerobic exercise maximum 3 sessions per week

Exclusion Criteria:

* Currently participating in an aerobic high intensity training program
* Smoker
* History of cardiovascular disease
* History of coronary heart disease
* Arrhythmias
* Heart failure/insufficiency
* Hypertension
* Diabetes
* Under medical treatment with anticoagulants, beta-blockers, calcium antagonists, bronchodilators, and/or steroids
* Psychological, neuromotor and/or osteo-muscular conditions that may affect participation in an exercise program.

Ages: 18 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in maximal oxygen uptake | Baseline and 8-weeks

SECONDARY OUTCOMES:
Change in systolic blood pressure | Baseline and 8-weeks
Change in diastolic blood pressure | Baseline and 8-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Víctor H Arboleda, MSc, Principal Investigator — Associate Professor; Elkin F Arango, MD. MSc, Principal Investigator — Associate Professor; Rubén D Gómez, PhD. MD, Principal Investigator — Professor; Yuri Feito, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Universidad de Antioquia, Medellín, Antioquia, Colombia

REFERENCES:
- [Derived] Arboleda-Serna VH, Feito Y, Patino-Villada FA, Vargas-Romero AV, Arango-Velez EF. Effects of high-intensity interval training compared to moderate-intensity continuous training on maximal oxygen consumption and blood pressure in healthy men: A randomized controlled trial. Biomedica. 2019 Sep 1;39(3):524-536. doi: 10.7705/biomedica.4451. PMID 31584766
- [Derived] Arboleda Serna VH, Arango Velez EF, Gomez Arias RD, Feito Y. Effects of a high-intensity interval training program versus a moderate-intensity continuous training program on maximal oxygen uptake and blood pressure in healthy adults: study protocol for a randomized controlled trial. Trials. 2016 Aug 18;17:413. doi: 10.1186/s13063-016-1522-y. PMID 27538896